CLINICAL TRIAL: NCT06893458
Title: Feeding Difficulties and Quality of Life in Children with Tracheal Cannula
Status: Not yet recruiting | Type: Observational
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Ida Engqvist, M.D, Karolinska Institutet
Other Study IDs: 2023-07493-01-IV
Record Dates: First submitted 2025-03-18; First posted 2025-03-25 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-01

CONDITIONS: Quality of Life (QOL); Tracheostomy; Children in the Pediatric Intensive Care Unit or General Pediatric Care Unit Requiring a Central Venous Catheter; Feeding Difficulties; Swallowing Difficulties; Caregiver Quality of Life
Keywords: pediatric quality of life; caregiver quality of life; swallowing related quality of life; feeding difficulties; pediatric tracheostomy
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Children with tracheostomy undergoing at LIVA: All children under 18 years with tracheostomy undergoing follow-up through the long term intensive care unit LIVA at Karolinska University Hospital Solna, Sweden will be eligible for inclusion. This is a majority of the children living with tracheostomy in Sweden.

SUMMARY:
The over all goal of this observational study is to study if there is an association between the presence of feeding difficulties and self-assessed quality of life in children with tracheal cannula.

The main questions it aims to answer are

1. What is the incidence of feeding difficulties in children with tracheostomy and what type of feeding difficulties affect these children?
2. How do children with a tracheal tube and their parents assess their quality of life measured through PedsQL?
3. Is there an association between the presence of feeding difficulties and self-assessed quality of life in children with tracheal cannula?

Quality of life will be assessed in an interview using the PedsQL instrument generic module 4.0. Swallowing difficulties will be assessed through evaluations based on The Montreal Children's Hospital Feeding Scale.

DETAILED DESCRIPTION:
Background:

Children with airway obstruction due to inborn malformations or trauma, or who have a chronic need for respiratory support due to lung- or neuromuscular diseases, may require a tracheostomy. A tracheostomy is a surgical opening of the trachea at the front of the neck to create an artificial airway, maintained with a tracheostomy tube. The Long-term Intensive Care Unit (LIVA) is a unit within Paediatric Perioperative Medicine and Intensive Care (BPMI) at Karolinska University Hospital. Since 1998, its primary task has been to care for children with tracheostomies from a large part of the country and it is the only unit of its kind in Scandinavia. LIVA's follow-up of children with tracheostomies includes regular team assessments and linked to LIVA is a multidisciplinary team consisting of paediatricians, ear-nose-throat specialists, paediatric anaesthesiologists, nurses, physiotherapists, dietitians, speech therapists, counsellors, and play therapists.

Studies indicate that feeding difficulties in children with tracheostomies are common and many have enteral feeding entirely or partially through gastrostomies. Our understanding regarding the types of feeding difficulties that these children experience and the potential causes and consequences however are limited. Studies have shown that both children and parents of children with tracheostomies rate their quality of life far lower than other groups of children with severe chronic diseases. Existing studies however are small involving only 20-25 subjects and studies of the quality of life of tracheostomized children in Sweden and the factors that may determine quality of life is lacking. A study in children with esophageal atresia indicate that the ability to taste food in the mouth is related to increased self assessed quality of life. The association between swallowing difficulties and quality of life in children with tracheostomy has to the best of our knowledge not been investigated before.

Main objective:

To investigate the quality of life in children with tracheostomy and their caregivers and identify the aspects determining it. Feeding difficulties will be studied specifically to investigate if there is an association between the ability to feed orally and self-assessed quality of life.

Research questions:

Primary: Is there an association between the presence of feeding difficulties and self-assessed quality of life in children with tracheal cannula? Secondary: How do children with a tracheal tube and their parents assess their quality of life measured through PedsQL? Which factors affect the quality of life in children with a tracheostomy?

Method: This is a prospective observational study. The 80 children currently undergoing regular follow-up at LIVA will be eligible for inclusion. Quality of life assessment by both children and parents is conducted using the PedsQL instrument, generic module 4.0. This validated tool is a questionnaire with 23 questions covering four domains: health/activities, emotions, social functioning, and school/daycare. Swallowing difficulties are assessed through evaluations based on The Montreal Children's Hospital Feeding Scale, a validated tool used to assess and monitor the feeding abilities and behaviors of infants and young children. Each assessment takes approximately 10min and will take place within the framework of the multidisciplinary team visits that the children associated with LIVA participate in.

Measures of quality of life are compared with data from other populations in the PedsQL database and related to the scores regarding feeding difficulties derived from the Montreal Feeding Scale.

Ethical approval has been obtained, ref. no 2023-07493-01.

ELIGIBILITY:
Inclusion Criteria: Children below the age of 18 with tracheostomy undergoing follow-up through the Long term Intensive Care Unit at Karolinska University Hospital in Stockholm Sweden between march 2025 and march 2027.

Exclusion criteria: Patients that can not undergo full evaluations/examinations will not be included.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children below the age of 18 with tracheostomy undergoing follow-up through the Long term Intensive Care Unit at Karolinska University Hospital in Stockholm Sweden between jan 2025 and jan 2027. About 80 patients.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-03-17 (Estimated); Primary Completion 2027-03-17 (Estimated); Study Completion 2027-03-17 (Estimated)

PRIMARY OUTCOMES:
Feeding difficulties in Children with Tracheostomy | 2 years
  Feeding difficulties are assessed based on The Montreal Children's Hospital Feeding Scale, a validated tool used to assess and monitor the feeding abilities and behaviors of infants and young children.
Quality of Life in children with Tracheostomy | 2 years
  Quality of life assessment by children with tracheostomy and their parents is conducted using the PedsQL instrument, generic module 4.0. This validated tool is a questionnaire with 23 questions covering four domains: health/activities, emotions, social functioning, and school/daycare.

SECONDARY OUTCOMES:
Association between Quality of life and presens of feeding difficulties | 2 years
  Measures of Quality of Life measures through PedsQl are related to the presens of feeding difficulty measured through the Montreal Childrens Hospital Feeding Scale.

CONTACTS AND LOCATIONS:
Locations (2):
- Sweden (2):
  - LIVA, Barn PMI, Karolinska Universitetssjukhuset Solna, Solna, Stockholm County
  - LIVA, Barn PMI, Karolinska Universitetssjukhuset, Solna, Sweden, Solna, Stockholm County

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Raynor EM, Wohl D. Tracheostomy-Related Swallowing Issues in Children. Otolaryngol Clin North Am. 2024 Aug;57(4):649-655. doi: 10.1016/j.otc.2024.02.017. Epub 2024 Mar 19. PMID 38508881
- [Background] Varni JW, Seid M, Kurtin PS. PedsQL 4.0: reliability and validity of the Pediatric Quality of Life Inventory version 4.0 generic core scales in healthy and patient populations. Med Care. 2001 Aug;39(8):800-12. doi: 10.1097/00005650-200108000-00006. PMID 11468499
- [Background] Ramsay M, Martel C, Porporino M, Zygmuntowicz C. The Montreal Children's Hospital Feeding Scale: A brief bilingual screening tool for identifying feeding problems. Paediatr Child Health. 2011 Mar;16(3):147-e17. doi: 10.1093/pch/16.3.147. PMID 22379377
- [Background] Varni JW, Limbers CA, Burwinkle TM. Impaired health-related quality of life in children and adolescents with chronic conditions: a comparative analysis of 10 disease clusters and 33 disease categories/severities utilizing the PedsQL 4.0 Generic Core Scales. Health Qual Life Outcomes. 2007 Jul 16;5:43. doi: 10.1186/1477-7525-5-43. PMID 17634123
- [Background] Bergmann S, Ritz LA, Widenmann-Grolig A, Jechalke S, von Schweinitz D, Hubertus J, Lurz E. Swallowing-related quality of life in children with oesophageal atresia: a national cohort study. Eur J Pediatr. 2023 Jan;182(1):275-283. doi: 10.1007/s00431-022-04677-4. Epub 2022 Nov 4. PMID 36331620
- [Background] Pullens B, Streppel M. Swallowing problems in children with a tracheostomy. Semin Pediatr Surg. 2021 Jun;30(3):151053. doi: 10.1016/j.sempedsurg.2021.151053. Epub 2021 May 21. PMID 34172203
- [Background] Henningfeld J, Lang C, Erato G, Silverman AH, Goday PS. Feeding Disorders in Children With Tracheostomy Tubes. Nutr Clin Pract. 2021 Jun;36(3):689-695. doi: 10.1002/ncp.10551. Epub 2020 Jul 23. PMID 32700397